CLINICAL TRIAL: NCT05517798
Title: Enamel Matrix Derivative for Alveolar Ridge Preservation After Tooth Extraction: a Randomized Controlled Trial
Brief Title: Enamel Matrix Derivative for Alveolar Ridge Preservation After Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Associate Professor Momen Atieh, Principal Investigator Associate Professor Momen Atieh, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBRUMHS
Record Dates: First submitted 2021-09-11; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Alveolar Ridge Preservation
Keywords: Alveolar ridge preservation; Dental implants; Enamel matrix derivative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xenograft + resorbable collagen membrane (Active Comparator): Bone grafting material (bovine origin) + resorbable collagen membrane (porcine origin)
  Interventions: Procedure: Alveolar ridge preservation
- Xenograft combined with EMD + resorbable collagen membrane (Active Comparator): Bone grafting material (bovine origin) with enamel matrix derivative (porcine origin) + resorbable collagen membrane (porcine origin)
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Alveolar ridge preservation is a method of decreasing bone resorption following tooth extraction and facilitating prosthetically-driven implant placement

SUMMARY:
The Global Burden of Disease Study of 2016 considered oral disease as the most common noncommunicable disease that affected half of the world population throughout their lifetime. Dental caries and periodontal diseases may cause pain and discomfort with severe forms of periodontal diseases causing tooth loss. Periodontal disease and tooth loss were estimated to be one of the ten causes of Years Lived with Disability. The dimensional changes in the alveolar ridge following tooth loss have been extensively investigated in the literature. At six months after tooth loss, a systematic review on bone remodelling showed horizontal and vertical bone loss of 29-63% and 11-22%, respectively. Such bone loss may complicate replacement of missing teeth with dental implants.

Dental implant is now a common treatment modality. However, the loss of bone volume may not allow the placement of dental implant in an optimal position and may subsequently jeopardize functional and aesthetic implant outcomes. Therefore, the use of bone replacement graft following tooth extraction, as part of a procedure termed alveolar ridge preservation (ARP), has increasingly becoming a common treatment protocol to optimize dental implant placement in the future.

A Cochrane review on ARP has demonstrated that there are no significant differences between the plethora of synthetic or biologically driven grafting materials used to minimize changes in width and height of the extraction sockets. Nevertheless, a regenerative agent, known as enamel matrix derivative (EMD), has gained more attention in regenerative therapy over the last 20 years. Several studies demonstrated its ability to enhance wound healing, induce new attachment and promote bone formation in recession and intrabony defects. Over the last two decades, EMD has been successfully used in the periodontal regeneration of intrabony defects. EMD has the potential to cause early vascularization and support early bone formation, hence, it can be considered as a potential regenerative agent for ARP when used with appropriate carrier material.

Moreover, the majority of studies showed that bone substitutes generally performed well in small or contained defects compared with non-grafted sites, but there is lack of information regarding the efficacy of different bone substitute materials in large defects. Short-term follow-up studies of three to six months have also dominated the literature when the main aim of the ARP is to develop a site that optimise long-term implant outcomes. Such aim requires evaluating the long-term performance of dental implants placed in preserved ridges and reporting patient outcomes in well-conducted randomized controlled trial.

The aim of the present clinical trial is to evaluate the adjunctive use of EMD in promoting the desired vascularization and bone fill in small and large defects following tooth extraction and report on the long-term implant and patient outcomes.

DETAILED DESCRIPTION:
A total of 34 participants, attending Dubai Dental Hospital, will be invited to take part in this randomized controlled trial. The participants will be randomly allocated to two equal sized groups (17 per group) using computer-generated numbers:

Control group (C): Xenograft (Bio-Oss Collagen, Geistlich Pharma AG, Wolhusen, Switzerland) + resorbable collagen membrane (Bio-Gide; Geistlich Pharma AG, Wolhusen, Switzerland).

Test group (T): Xenograft (Bio-Oss Collagen, Geistlich Pharma AG, Switzerland) combined with EMD (Straumann Emdogain, Straumann AG, Basel, Switzerland) + resorbable collagen membrane (Bio-Gide; Geistlich Pharma AG, Wolhusen, Switzerland). The minimally traumatic extraction of the tooth will include raising a full mucoperiosteal flap and sectioning the roots if required. This will allow visual assessment of the socket walls and thorough debridement of the extraction socket. A clinician not involved in the study will then open a sealed opaque envelope and ARP procedure will be carried out by placing either xenograft (Bio-Oss Collagen, Geistlich Pharma AG, Switzerland) alone or combined with EMD (Straumann Emdogain, Straumann AG, Basel, Switzerland). The xenograft (Bio-Oss Collagen, Geistlich Pharma AG, Switzerland) will pre-wetted with blood or saliva prior to applying it to the socket. EMD (Straumann Emdogain, Straumann AG, Basel, Switzerland) will then be placed into the socket. Xenograft will not be mized with EMD outside the oral cavity. In both groups, a resorbable collagen membrane (Bio-Gide; Geistlich Pharma AG, Wolhusen, Switzerland) will be trimmed and adapted to cover the socket. The flaps will then be replaced and sutured with 4/0 polyglycolic acid interrupted and mattress sutures.

After six months of healing, CBCT will be utilized in the assessment of the available bone volume and virtual implant treatment planning. A three-dimensional printed surgical stent will be fabricated to aid in implant placement. The implant site will then be prepared according to the surgical protocol outlined in the International Team for Implantology (ITI) consensus conference. This procedure will include raising a mucoperiosteal flap with slightly palatal crestal incision and sulcular incision extending to the adjacent teeth. The osteotomy will be prepared to place a chemically modified, sand-blasted and acid-etched dental implants. In the presence of peri-implant bone defect, simultaneous contour augmentation will be carried out. For all implant surgeries, two-stage protocol will be followed with a re-opening procedure after 12 weeks to place a healing abutment.

Prosthodontic Protocol The restorative phase will be carried out in a partial or complete digital workflow. Within 21-28 days of placing the healing abutment, the implant position will be captured using an intraoral optical scanner. Computer-aided design / computer-aided manufacturing (CAD/CAM) will be utilizing the captured digital data to design a screw-retained crown, which will then be milled of monolithic lithium disilicate blanks and bonded to pre-fabricated titanium abutments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Require extraction of anterior or posterior single tooth due to caries, endodontic and prosthetic complications.
* The tooth that requires extraction is bordered by two teeth.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline).
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Localised / generalised periodontitis.
* Presence of acute periapical lesion.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* Long term use of non-steroidal anti-inflammatory medications.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Severe bruxism or parafunctional habits.
* Large occlusal discrepancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival / success rate after one year | 1 year
  'Implant survival' means that implants are still in the mouth at the time of examination
Patient postoperative experience | 1 week
  Postoperative experience means any events occurring after and relating to the procedure
Implant survival / success rate after two years | 2 years
  'Implant survival' means that implants are still in the mouth at the time of examination
Implant survival / success rate after three years | 3 years
  'Implant survival' means that implants are still in the mouth at the time of examination

SECONDARY OUTCOMES:
Changes in width and height of alveolar ridge | 6 months
  Differences in bony dimensions before and after alveolar ridge preservation, meaasured in millimeters using cone beam computed tomography
Bone quality | 1 day
  Bone quality relates to the degree of bone density present
Need for additional bone augmentation | 1 day
  Since all the sites had alveolar ridge preservation, we would like to assess whether another bone grafting is required at the time of placing implants. The assessment is YES or NO and it is only assessed ONE TIME ... AT THE TIME OF IMPLANT PLACEMENT
Changes in peri-implant marginal bone level | 1 year
  Differences in level of bone surrounding the implant

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No